CLINICAL TRIAL: NCT01190800
Title: Decision Capacity Assessment in Persons With Alzheimer's Disease: Approach by Capacity to Appoint a Proxy, to Consent to Treatment and to Vote
Brief Title: Capacity Assessment in Persons With Alzheimer's Disease
Acronym: MACAP
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: NI 08009
Record Dates: First submitted 2010-08-27; First posted 2010-08-30 (Estimated); Last update posted 2014-10-15 (Estimated); Status verified 2014-06

CONDITIONS: Alzheimer's Disease; Capacity to Consent to Treatment; Capacity to Vote; Capacity to Design a Proxy
Keywords: Alzheimer's Disease; Capacity assessment; Decision-making assessment; Capacity to consent to treatment; Capacity to vote; Capacity to appoint a proxy
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Biospecimen Retention: None Retained — None Retained
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to assess decision-making capacity in persons with Alzheimer's disease. First, our goal is to validate four French capacity assessment tools for persons with Alzheimer's Disease : a French version of the Competency Assessment Tool for Consent to Treatment and of the Competency Assessment Tool for Voting, two questionnaires assessing the capacity to appoint a proxy either to consent to treatment or to vote. Second, once validated, we plan these questionnaires to study decision-making abilities and their determinants in persons with Alzheimer's disease and control subjects.

DETAILED DESCRIPTION:
Study of Alzheimer's disease patients show a wide variability in decision-making abilities, especially for the consent to treatment and the ability to vote. No tools are available to assess the capacity to design a proxy. The purpose of this research is to assess simultaneously four decision-making abilities in persons with Alzheimer's disease: the capacity to consent to treatment, the capacity to vote and the capacity to design a proxy either to consent to treatment or to vote.

This study will recruit 320 patients with Alzheimer's disease and 80 non-demented control subjects. Four decision-making questionnaires will be administered to participants to explore participant capacity to understand, reason, appreciate and make a choice about the capacity to consent to treatment, to vote and to design a proxy either to consent to treatment or to vote. Once validated in the first part of this research, the questionnaires will be used to study decision-making abilities and their determinants in patients with Alzheimer's disease and control subjects.

ELIGIBILITY:
Inclusion Criteria:

* for patients with Alzheimer's disease: age >=18 years, to be native speakers of French and French nationality, Diagnosed with a Alzheimer's disease and followed in a French "Centre Memory of Resources and Research"(CMRR)
* for control subjects: age >=18 years, to be native speakers of French and French nationality, have no complaints of memory problems, primary caregiver of patient with AD of the same age as the patient nearly 10 years

Exclusion Criteria:

* for all participants: confusion, severe psychiatric disorders, stroke, blindness, uncorrected hearing loss, refusal to participate in the study
* for patients with Alzheimer's disease: other dementia than AD
* for control subjects: diagnosed dementia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: persons with Alzheimer's disease
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2010-06; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Antoine Bosquet, MD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Hôpital Louis Mourier, Colombes, France